CLINICAL TRIAL: NCT06906991
Title: Psychological Treatment Based on the Unified Protocol for Emotional Regulation in Individuals With Fibromyalgia: What Does It Add to the Multicomponent FIBROWALK Therapy? A Randomized Controlled Trial
Brief Title: Multicomponent FIBROWALK Therapy Plus Unified Protocol for Emotional Regulation in Individuals With Fibromyalgia
Acronym: FIBROWALK+UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBROWALK+UP
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia (FM)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial (RCT) with two intervention groups: (1) FIBROWALK only and (2) FIBROWALK + Unified Protocol (UP). Participants will be assessed at baseline (pre-treatment), post-treatment, and at a six-month follow-up. The study will enroll 182 participants with fibromyalgia, based on eligibility criteria set by the Rheumatology Service at Vall d'Hebron Hospital.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIBROWALK Program (Active Comparator): Multicomponent group-based therapy including therapeutic exercise, pain neuroscience education, CBT, and mindfulness.
  Delivered over 12 weekly group sessions (2 hours per session).
  Interventions: Behavioral: FIBROWALK
- FIBROWALK + Unified Protocol (UP) (Experimental): Participants receive the same FIBROWALK intervention, plus the Unified Protocol (UP), a psychological transdiagnostic intervention which will be delivered individually in parallel.
  The UP consists of 12 individual sessions (50-60 minutes each), covering modules on emotional awareness, distress tolerance, and reducing avoidance.
  Interventions: Behavioral: FIBROWALK; Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: FIBROWALK — FIBROWALK is a structured, multicomponent therapeutic program designed specifically for patients with fibromyalgia, combining evidence-based interventions that target both physical and emotional symptoms of the condition. Unlike traditional standalone interventions (e.g., exercise-only or CBT-only), FIBROWALK integrates multiple therapeutic modalities in a holistic, group-based format to address the broad symptom profile of fibromyalgia, including chronic pain, fatigue, and impaired functionality. Sessions are delivered in groups of up to 20 participants, fostering peer support and shared learning.
  Key Components of FIBROWALK:
  * Therapeutic Exercise
  * Pain Neuroscience Education
  * Cognitive-Behavioral Therapy
  * Mindfulness-Based Stress Reduction
  * Psychoeducation
Behavioral: Unified Protocol — The Unified Protocol (UP) is a transdiagnostic, cognitive-behavioral therapy (CBT) intervention designed to address emotional dysregulation across a range of mental health conditions. Unlike traditional disorder-specific CBT interventions (e.g., CBT for anxiety or depression), the UP targets core emotional processes common to multiple disorders, making it particularly suitable for fibromyalgia patients who often experience comorbid anxiety, depression, and emotional distress. Unlike condition-specific therapies, the UP addresses the shared emotional mechanisms underlying anxiety, depression, and chronic pain, making it well-suited for fibromyalgia patients with complex emotional and physical symptomatology. UP emphasizes increasing tolerance to emotional and physical discomfort, a critical area for fibromyalgia patients who often experience heightened emotional reactivity and pain sensitivity.
  The UP is delivered individually and consists of 12 structured, manualized modules.
  Arms: FIBROWALK + Unified Protocol (UP)

SUMMARY:
Fibromyalgia is a chronic condition characterized by widespread pain, fatigue, sleep disturbances, and cognitive dysfunction. Although the FIBROWALK multicomponent program improves physical functionality and pain, its impact on emotional regulation remains limited. This study aims to integrate the Unified Protocol (UP), a cognitive-behavioral therapy (CBT) approach, to enhance emotional and physical distress tolerance in fibromyalgia patients and explore participants' satisfaction, difficulties, and barriers to treatment.

This study investigates the efficacy of integrating the Unified Protocol (UP), a transdiagnostic intervention based on CBT, with the multicomponent FIBROWALK therapy for individuals with fibromyalgia. The trial seeks to enhance emotional regulation, reduce anxiety and depression, and improve quality of life. Additionally, it will gather qualitative feedback from participants to identify challenges, barriers, and potential improvements to the therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with fibromyalgia, according to the 2011 American College of Rheumatology (ACR) modified criteria.
* Aged 18 or older.

Exclusion Criteria:

* Individuals with psychotic disorders, substance abuse, or severe cognitive impairment (based on medical evaluation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up. Changes in anxiety and depression scores from baseline to post-treatment and 6-month follow-up.
  This scale will measure changes in anxiety and depression levels. HADS is a validated 14-item questionnaire specifically designed to detect anxiety and depression symptoms in patients with chronic health conditions, including fibromyalgia.
Fibromyalgia Impact Questionnaire - Revised (FIQ-R) | Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up. Changes in functioning scores from baseline to post-treatment and 6-month follow-up.
  This tool will assess the overall impact of fibromyalgia on patients' daily functionality, covering physical limitations, pain intensity, fatigue, and general well-being. Higher scores indicate worse fibromyalgia impact.

SECONDARY OUTCOMES:
Frustration Discomfort Scale (FDS) | Changes in distress tolerance scores from baseline to post-treatment and 6-month follow-up. Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up.
  This questionnaire evaluates participants' tolerance to frustration and emotional distress, which are key targets in the Unified Protocol intervention. It measures responses to challenging emotional and physical experiences.
Satisfaction with Life Scale (SWLS) | Changes in satisfaction with life scores from baseline to post-treatment and 6-month follow-up. Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up.
  This scale measures participants' subjective well-being and overall life satisfaction. It consists of five items that assess life satisfaction on a 7-point Likert scale.
Visual Analog Scales (VAS) for Pain and Fatigue | Changes in pain and fatigue scores from baseline to post-treatment and 6-month follow-up. Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up.
  Self-reported scales ranging from 0 (no pain/fatigue) to 10 (worst possible pain/fatigue) will be used to assess the perceived intensity of pain and fatigue, which are core symptoms of fibromyalgia.
Psychological Inflexibility in Pain Scale (PIPS) | Changes in psychological inflexibility scores from baseline to post-treatment and 6-month follow-up. Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up.
  This scale measures two key factors in chronic pain patients: cognitive fusion (difficulty detaching from pain-related thoughts) and experiential avoidance (efforts to avoid or control pain-related experiences).
Credibility/Expectancy Questionnaire (CEQ) | Changes in perceived credibility of and expectations for the treatment scores from baseline to post-treatment. Administered at baseline and post-treatment (12 weeks).
  This 6-item questionnaire assesses participants' perceived credibility of and expectations for the treatment. It will be administered both at baseline to measure initial expectations and post-treatment to measure changes in perception.
Blood Neutrophil-Lymphocyte Ratio (NLR) | Changes in NLR scores from baseline to post-treatment and 6-month follow-up. Baseline (pre-treatment), post-treatment (12 weeks), and at 6-month follow-up.
  The neutrophil-lymphocyte ratio (NLR) will be measured as a marker of systemic inflammation. NLR has been associated with inflammatory responses in various chronic conditions, including fibromyalgia. This ratio will be calculated by dividing the absolute neutrophil count by the absolute lymphocyte count from blood samples collected at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Vall Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
At this time, the individual participant data (IPD) collected during the study will not be shared publicly due to privacy concerns and the ethical requirements related to handling sensitive health data. The study follows GDPR (General Data Protection Regulation) and Spanish national regulations (LOPD 3/2018) on the protection and confidentiality of personal health information.
  Although the data will be anonymized and securely stored, sharing IPD outside the research team may not be feasible without additional participant consent and institutional approvals. Requests for data access may be considered on a case-by-case basis and must align with ethical guidelines, institutional policies, and data protection laws.

REFERENCES:
- [Background] Serrat M, Sanabria-Mazo JP, Almirall M, Muste M, Feliu-Soler A, Mendez-Ulrich JL, Sanz A, Luciano JV. Effectiveness of a Multicomponent Treatment Based on Pain Neuroscience Education, Therapeutic Exercise, Cognitive Behavioral Therapy, and Mindfulness in Patients With Fibromyalgia (FIBROWALK Study): A Randomized Controlled Trial. Phys Ther. 2021 Dec 1;101(12):pzab200. doi: 10.1093/ptj/pzab200. PMID 34499174
- [Background] Serrat M, Coll-Omana M, Albajes K, Sole S, Almirall M, Luciano JV, Feliu-Soler A. Efficacy of the FIBROWALK Multicomponent Program Moved to a Virtual Setting for Patients with Fibromyalgia during the COVID-19 Pandemic: A Proof-of-Concept RCT Performed Alongside the State of Alarm in Spain. Int J Environ Res Public Health. 2021 Sep 30;18(19):10300. doi: 10.3390/ijerph181910300. PMID 34639600
- [Background] Suso-Ribera C, Camacho-Guerrero L, Osma J, Suso-Vergara S, Gallardo-Pujol D. A Reduction in Pain Intensity Is More Strongly Associated With Improved Physical Functioning in Frustration Tolerant Individuals: A Longitudinal Moderation Study in Chronic Pain Patients. Front Psychol. 2019 Apr 26;10:907. doi: 10.3389/fpsyg.2019.00907. eCollection 2019. PMID 31133917
- [Background] Osma J, Martinez-Garcia L, Quilez-Orden A, Peris-Baquero O. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Medical Conditions: A Systematic Review. Int J Environ Res Public Health. 2021 May 11;18(10):5077. doi: 10.3390/ijerph18105077. PMID 34064898
- [Background] Barlow, D. H., Farchione, T. J., Sauer-Zavala, S., Latin, H. M., Burris, J. R., Bentley, K. H., Boettcher, H. T., & Cassiello-Robbins, C. (2019). Protocolo unificado para el tratamiento transdiagnóstico de los trastornos emocionales: Manual del terapeuta (J. J. Osma López & E. Crespo Delgado, Trads.; Segunda edición revisada y actualizada). Alianza Editorial.
- [Background] Angarita-Osorio N, Perez-Aranda A, Feliu-Soler A, Andres-Rodriguez L, Borras X, Suso-Ribera C, Slim M, Herrera-Mercadal P, Fernandez-Vergel R, Blanco ME, Luciano JV. Patients With Fibromyalgia Reporting Severe Pain but Low Impact of the Syndrome: Clinical and Pain-Related Cognitive Features. Pain Pract. 2020 Mar;20(3):255-261. doi: 10.1111/papr.12847. Epub 2019 Nov 11. PMID 31627253
- [Background] Allen LB, Tsao JCI, Seidman LC, Ehrenreich-May J, Zeltzer LK. A Unified, Transdiagnostic Treatment for Adolescents With Chronic Pain and Comorbid Anxiety and Depression. Cogn Behav Pract. 2012 Feb;19(1):56-67. doi: 10.1016/j.cbpra.2011.04.007. PMID 28824271